CLINICAL TRIAL: NCT01958762
Title: Screening for Cancers in the Oral CAvity Targeting Tobacco Users in Somme, France
Brief Title: Screening for Cancers in the Oral CAvity
Acronym: IDECAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Picardy - Regional health agency (ARS) (Unknown); Regional Council Picardie (Unknown); Regional Observatory of Health and Social Issues in Picardie (OR2S) (Unknown); Association for the screening of diseases in Somme (Adema 80) (Unknown); Somme Cancer Registry (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI2013_843_0010; 2013-A00606-39 (Other: ID-RCB)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Oral Cavity Cancer
Keywords: Screening; Cancer; Tobacco; General Practitioner; Precancerous Lesion; Dysplasia; Tobacco vendor
MeSH Terms: conditions — Mouth Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Screening for cancers in the oral cavity (Other)
  Interventions: Other: Invitation for oral cavity cancer screening

INTERVENTIONS:
Other: Invitation for oral cavity cancer screening

SUMMARY:
In the Somme region of France, cancer registry data showed an increasing incidence of oral cancer. The Incidence Rates in Somme as compared to the national rates for Lip, Oral Cavity and Pharynx Cancer were in 2010: 31,4/100 000 Standard population versus 18,2 /100 000 for male and 8,2/100 000 versus 5,5/100 000 for female, disaster area where action to improve early detection for smokers will be assessed. This target population consults late (as 70% of oral cavity cancers are diagnosed at a late stage (T3 or T4). This project is an innovative incentive strategy for screening among general practitioners based on unusual information vectors (tobacconist, local media).

The main objective of this study is a screening of oral cavity cancers in tobacco users aged 30-75 years in the Somme region of France.

DETAILED DESCRIPTION:
Methodology:

* Education and alerting physicians to the early detection of cancers of oral cavity and coordination of networks involved for 1 year.
* Incentive period for the screening by the tobacconist who distributes with every package of cigarettes bought a flyer of invitation to the screening.
* Carrying out screening examinations by general practitioners with completion of the customized examination forms, orientation towards a specialist, data collection and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Any smoker who buys a pack of cigarettes over a period of two weeks in a tobacco shop located on the territory of the Somme
* lives in somme departement

Exclusion Criteria:

-

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Participation rate to the screening of the target patients. | 03 months after the start of the incentive period
  Numbers of people who benefit from a screening exam by a physician of the Somme region in comparison, with the target population of the Somme region. This rate will be also calculated according the different of age and sex.

SECONDARY OUTCOMES:
The participation rate of the physicians. | 03 months after the start of the incentive period
  Number of physicians who send back at least one clinical form compared to the numbers of physician of the Somme.
The participation rate of the tobacco venders. | 15 days after the start of the incentive period
  The number of tobacco venders who gave at least 01 " Flyer " in comparison to the numbers of tobacco venders of the Somme.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DEVAUCHELLE, MD, phD, Principal Investigator — Amiens University Hospital
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

REFERENCES:
- [Background] http://www.cepidc.vesinet.inserm.fr/
- [Background] Bailey EE, Marghoob AA, Orengo IF, Testa MA, White VR, Geller AC. Skin cancer knowledge, attitudes, and behaviors in the salon: a survey of working hair professionals in Houston, Texas. Arch Dermatol. 2011 Oct;147(10):1159-65. doi: 10.1001/archdermatol.2011.184. PMID 22006132
- [Background] Subramanian S, Sankaranarayanan R, Bapat B, Somanathan T, Thomas G, Mathew B, Vinoda J, Ramadas K. Cost-effectiveness of oral cancer screening: results from a cluster randomized controlled trial in India. Bull World Health Organ. 2009 Mar;87(3):200-6. doi: 10.2471/blt.08.053231. PMID 19377716
- [Background] Epstein JB, Silverman S Jr, Epstein JD, Lonky SA, Bride MA. Analysis of oral lesion biopsies identified and evaluated by visual examination, chemiluminescence and toluidine blue. Oral Oncol. 2008 Jun;44(6):538-44. doi: 10.1016/j.oraloncology.2007.08.011. Epub 2007 Nov 8. PMID 17996486
- [Background] Hubert A, Lapôtre B, Raverdy N, Ganry O. Incidence et mortalité 2002-2004 Evolution de 1982 à 2004. Registre du Cancer de la Somme. Juin 2009. 138 p.
- [Background] Réseau Francim, service de biostatistique des hospices civils de Lyon. Survie des patients atteints de Cancer en France : étude des registres du réseau Francim, Paris 2007, springer, 406
- [Background] Reyt E, Righini C. Les cancers du plancher buccal. La chirurgie mini-invasive. Société française de carcinologie cervico-faciale.EDK